CLINICAL TRIAL: NCT03329105
Title: Efficacy of a Rinse Containing Sea Salt and Lysozyme on Biofilm and Gingival Health in a Group of Young Adults: A Pilot Study.
Brief Title: Efficacy of a Rinse Containing Sea Salt and Lysozyme on Biofilm and Gingival Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jay Hoover, Principal Investigator, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-272
Record Dates: First submitted 2017-10-17; First posted 2017-11-01 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Chronic Gingivitis; Chronic Gingivitis, Plaque Induced
Keywords: Gingival Health; Biofilm Formation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sea Salt Mouth Rinse (Experimental)
  Interventions: Other: Sea Salt Mouth Rinse; Other: Standardized Oral Health Practices
- Standardized Oral Health Practices (Active Comparator)
  Interventions: Other: Standardized Oral Health Practices

INTERVENTIONS:
Other: Sea Salt Mouth Rinse — Rinsing mouth with a tablespoon of sea salt mouth rinse without any dilution, for 30 seconds, once in the morning and once before bed, in addition to Standardized Oral Health Practices.
  Arms: Sea Salt Mouth Rinse
Other: Standardized Oral Health Practices — Brushing teeth for two minutes using the modified Bass technique, twice per day with the provided dentifrice, and flossing once daily using the spool method

SUMMARY:
This study evaluates the addition of a mouth rinse containing sea salt, xylitol and lysozyme to standardized oral health practices on biofilm formation and gingival health in a group of young adults.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a new sea salt mouth rinse containing xylitol and the antibacterial enzyme, lysozyme on biofilm formation and gingival health in a group of young adults. Xylitol is a well-established non-sugar sweetener and an anti-caries agent. The use of this polyol results in loosely adherent biofilms by reducing the amount of extracellular lipopolysaccharides and lipoteichoic acids, facilitating its easy removal by mechanical means. Lysozymes are antibacterial proteins that hydrolyze the linkage between N-acetylmuramic acid and N-acetylglucosamine of peptidoglycan in the cell wall of Gram + bacteria effectively limiting growth.

ELIGIBILITY:
Inclusion Criteria:

* Dentate
* Medically healthy
* No orthodontic bands
* An anticipated ability to attend the two scheduled visits

Exclusion Criteria:

* Significant medical condition (including but not limited to, poorly controlled diabetes mellitus, rheumatic heart disease or clinically significant heart murmur)
* Pregnancy
* Recent history of, or ongoing, antibiotic therapy

Ages: 20 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
Turesky modification of Quigley-Hein plaque index | Change from Baseline at 1 Month
  Evaluation of plaque scores on six representative teeth: 16, 21, 24, 36, 41 & 44, using an index that evaluates the plaque revealed on the buccal and lingual non-restored surfaces of the teeth on a scale of 0 to 5, defined by G. A. Quigley and J. W. Hein in 1962 and modified by S. Turesky, N. D. Gilmore, and I. Glickman in 1970.
Presence or absence of gingival bleeding | Baseline and 1 Month
  Presence or absence of gingival bleeding on gentle probing to determine gingival health

CONTACTS AND LOCATIONS:
Overall Officials: Jay Hoover, Principal Investigator — Professor, College of Dentistry
Locations (1):
- College of Dentistry, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albandar JM, Rams TE. Global epidemiology of periodontal diseases: an overview. Periodontol 2000. 2002;29:7-10. doi: 10.1034/j.1600-0757.2002.290101.x. No abstract available. PMID 12102700
- [Background] Burt B; Research, Science and Therapy Committee of the American Academy of Periodontology. Position paper: epidemiology of periodontal diseases. J Periodontol. 2005 Aug;76(8):1406-19. doi: 10.1902/jop.2005.76.8.1406. No abstract available. PMID 16101377
- [Background] Axelsson P, Lindhe J, Nystrom B. On the prevention of caries and periodontal disease. Results of a 15-year longitudinal study in adults. J Clin Periodontol. 1991 Mar;18(3):182-9. doi: 10.1111/j.1600-051x.1991.tb01131.x. PMID 2061418
- [Background] Bizarra F, Ribeiro S. Improving toothbrushing behaviour in an institution for the disabled in Lisbon, Portugal. Int J Dent Hyg. 2009 Aug;7(3):182-7. doi: 10.1111/j.1601-5037.2009.00387.x. PMID 19659714
- [Background] Litonjua LA, Cabanilla LL, Abbott LJ. Plaque formation and marginal gingivitis associated with restorative materials. Compend Contin Educ Dent. 2011 May;32(4):e69-72. PMID 23738894
- [Background] Brecx M. Strategies and agents in supragingival chemical plaque control. Periodontol 2000. 1997 Oct;15:100-8. doi: 10.1111/j.1600-0757.1997.tb00109.x. No abstract available. PMID 9643237
- [Background] Jackson RJ. Metal salts, essential oils and phenols--old or new? Periodontol 2000. 1997 Oct;15:63-73. doi: 10.1111/j.1600-0757.1997.tb00106.x. No abstract available. PMID 9643234